CLINICAL TRIAL: NCT04499469
Title: The Role of Spreader Grafts in Reduction Rhinoseptoplasty: a Randomized Clinical Trial With Quality of Life Assessment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 91672218400005327
Record Dates: First submitted 2020-07-21; First posted 2020-08-05 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-07

CONDITIONS: Rhinoplasty; Nasal Obstruction
MeSH Terms: conditions — Nasal Obstruction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spreader Graft (Experimental): Placement and attachment with 5.0 polydioxanone (PDS) suture 2 grafts in the middle third of the nose
  Interventions: Procedure: Spreader Graft
- Without Spreader Graft (No Intervention): No engraftment in the middle third

INTERVENTIONS:
Procedure: Spreader Graft — To place and attach with 5.0 PDS suture 2 grafts in the middle third of the nose
  Other Names: Middle Third Grafts
  Arms: Spreader Graft

SUMMARY:
Nasal obstruction is one of the majors concerns in reduction rhinoseptoplasty, because it affects quality of life and surgical outcomes. Is the association of middle third grafts with reduction rhinoseptoplasty responsible for an increase in quality of life related to nasal obstruction when compared to reduction rhinoseptoplasty without the placement of these grafts?

DETAILED DESCRIPTION:
Reduction rhinoplasty and rhinoseptoplasty are among the most accomplished aesthetic procedures in Plastic Surgery and Otorhinolaryngology. Nasal obstruction is one of the majors concerns in this procedures, because it affects quality of life and surgical outcomes. Nasal surgeons have paid much attention to nasal valve area to prevent nasal obstruction and some assert reconstruction of the middle vault after dorsal reduction with grafts. The gold standard for middle vault reconstruction after dorsal reduction has been the spreader graft, first advocated by Sheen. Studies in surgical techniques for the treatment of nasal valve collapse focus much more in techniques than in evidence of its efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for reduction rhinoseptoplasty who agreed to participate in the study and who did not meet the exclusion criteria

Exclusion Criteria:

* Absence of nasal obstruction;
* Previous nasosinusal surgery;
* Symmetrical or asymmetric insufficiency of the middle third that would justify the placement of middle third grafts for the treatment of these problems;
* Presence of nasal valve insufficiency as the only cause of nasal obstruction;
* Cranio-facial anomalies;
* Presence of nasosinusal tumors;
* Active acute rhinosinusitis;
* Patients undergoing treatment of other entities concomitant to rhinoseptoplasty such as: sinus inflammatory surgery, adenoid hypertrophy removal, septal perforation correction, otoplasty or blepharoplasty.

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-10-03 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Nasal Obstruction Symptom Evaluation Scale (NOSE) | 180 postoperative days
  The NOSE will be used to measure the quality of life related to nasal obstruction. It is a validated instrument specifically designed for use in patients with nasal obstruction. According to this scale patients are asked to evaluate difficulty breathing in a general way and specifically the difficulty in breathing through the nose, breathing during sleep, and severity of their nasal congestion. The severity of the symptoms is recorded on a scale of 0 to 4, with 0 being the absence of a problem and 4 being a serious problem. The possible scores range from 0 to 20 and the higher scores indicate a higher degree of nasal obstruction. The sum of the scores is multiplied by 5 so as to obtain a final score ranging from 0 to 100, with higher values associated with poorer quality of life.
  The scale will be applied at the base line and at 30, 90 and 180 postoperative days.

SECONDARY OUTCOMES:
Rhinoplasty Outcome Evaluation (ROE) Scale | 180 postoperative days
  The ROE scale is a questionnaire, designed for the evaluation of rhinoplasty results. This instrument is composed of six questions that assess three domains of quality of life: physical, mental / emotional and social. Each question is scored on a scale of 0 to 4 and converted to a total score of 0 to 100, dividing the value by 24 and multiplying by 100. A score above 85 is considered excellent and generally means that the patient is very satisfied. However, the comparison of pre and postoperative values usually provide the most relevant information. Patients will be asked to respond to this scale in the base line and at 30, 90 and 180 postoperative days.
Visual Analogue Scale - Nasal Obstruction | 180 postoperative days
  Patients will be asked to complete an analogue-visual scale indicating the degree of nasal obstruction, with the instrument Visual Analogue Scale (VAS). The VAS for nasal obstruction has 100 mm and this scale will be converted into a scale ranging from 0 to 100, and the value "0" represents no nasal obstruction and the value "100" correspond to the highest nasal obstruction level possible. The scale will be applied in the base line as well as in the 30,90 and 180 postoperative days.
Clinical Diagnosis of Allergic Rhinitis | Base line and 180 postoperative days
  A questionnaire of symptoms and intensity based in Allergic Rhinitis and its Impact on Asthma (ARIA) recommendations and treatment of Allergic Rhinitis is applied in the base line and 30, 90 and 180 postoperative days
Complications | 7 until 180 postoperative days
  The protocol includes data such as bleeding, signs of graft detachment, presence of crusts, residual septal deviation, synechiae and septal perforation to be to be evaluated on the 7th, 30th, 90th and 180th postoperative days
Anterior Rhinoscopy and Nasal Endoscopy | Base line and 180 postoperative days
  All patients will be submitted to anterior rhinoscopy and nasal endoscopy using a 0 degree rigid nasal endoscope. The septal deviation will be classified considering the side of maximum deviation (right / left), the severity of the obstruction caused by the septal deviation (<25% of obstruction, 25-50% of obstruction, 50-75% of obstruction;> 75% of obstruction) and the location of the point of greatest deviation based on the classification of the five Cottle areas.
  The evaluation of this outcome will be performed in the preoperative consultation, 30, 90 and 180 after the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Lavinsky-Wolff, PhD, Study Director — Federal University of Health Science of Porto Alegre
Locations (1):
- Raphaella Migliavacca, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided